CLINICAL TRIAL: NCT06676904
Title: Neonatal Platelet Transfusion Threshold Trial
Acronym: NeoPlaTT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NICHD-NRN-0065; 1U24HL173304-01 (NIH); UG3HL173303 (NIH)
Record Dates: First submitted 2024-10-03; First posted 2024-11-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Thrombocytopenia; Neonatal; Platelet Transfusion; Infant, Newborn, Diseases; Infant, Extremely Low Birth Weight; Infant, Small for Gestational Age; Thrombosis
Keywords: platelet transfusion; neonatal; thrombosis
MeSH Terms: conditions — Thrombocytopenia; Infant, Newborn, Diseases; Thrombosis

STUDY DESIGN:
Intervention Model Description: Randomized trial with 1:1 allocation to parallel arms within strata of Study Center and gestational age (23-24 weeks and 25-26 weeks PMA). Multiples will be randomized independently. Approximately 30% of enrolled participants are expected to meet the platelet count threshold for randomization. The target sample size for randomization is 730, or 365 per arm.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: There will be no blinding/masking of the treatment group allocation to providers or parents to ensure providers are aware of treatment allocation to guide platelet transfusions. This is necessary to ensure adherence to the treatment arms. However, a standard tool will be used to assess bleeding as described below and grading of the severity of bleeding will be performed centrally. In addition, radiologists interpreting cranial ultrasound findings will be blinded to treatment arm allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher Platelet Transfusion Threshold (Active Comparator): Infants randomized to this arm will be monitored for a platelet transfusion threshold of 50 x 10^9/L during postnatal days 1-7, and then for a platelet transfusion threshold of 35 x 10^9/L at 8 or more postnatal days of life. Infants will remain on this protocol-driven threshold through 40 0/7 weeks postmenstrual age. The platelet dose will be 10 ml/kg administered over 60-120 minutes.
  Interventions: Procedure: Higher Platelet Transfusion Threshold
- Lower Platelet Transfusion Threshold (Other): Infants randomized to this arm will be monitored for a platelet transfusion threshold of 25 x 10^9/L during postnatal days 1-7, and then for a platelet transfusion threshold of 20 x 10^9/L at 8 or more postnatal days of life. Infants will remain on this protocol-driven threshold through 40 0/7 weeks postmenstrual age. The platelet dose will be 10 ml/kg administered over 60-120 minutes.
  Interventions: Procedure: Lower Platelet Transfusion Threshold

INTERVENTIONS:
Procedure: Higher Platelet Transfusion Threshold — Infants randomized to this arm will be monitored for a platelet transfusion threshold of 50 x 10^9/L during postnatal days 1-7, and then for a platelet transfusion threshold of 35 x 10^9/L at 8 or more postnatal days of life. Infants will remain on this protocol-driven threshold through 40 0/7 weeks postmenstrual age. The platelet dose will be 10 ml/kg administered over 60-120 minutes.
  Other Names: Liberal Transfusion Threshold
  Arms: Higher Platelet Transfusion Threshold
Procedure: Lower Platelet Transfusion Threshold — Infants randomized to this arm will be monitored for a platelet transfusion threshold of 25 x 10^9/L during postnatal days 1-7, and then for a platelet transfusion threshold of 20 x 10^9/L at 8 or more postnatal days of life. Infants will remain on this protocol-driven threshold through 40 0/7 weeks postmenstrual age. The platelet dose will be 10 ml/kg administered over 60-120 minutes.
  Other Names: Restrictive Transfusion Threshold
  Arms: Lower Platelet Transfusion Threshold

SUMMARY:
The objective of the NeoPlaTT trial is to test whether, among extremely preterm infants born at 23 0/7 to 26 6/7 weeks' gestation, a lower platelet transfusion threshold, compared to a higher threshold, improves survival without major or severe bleeding up to 40 0/7 weeks' postmenstrual age (PMA).

DETAILED DESCRIPTION:
Thrombocytopenia, defined as a platelet count <150 x 10^9/L, is a common neonatal problem that affects 22% to 35% of infants admitted to the neonatal intensive care unit. Platelets are important for primary hemostasis to prevent blood extravasation after vascular injury. Based on the role of platelets in hemostasis, prophylactic platelet transfusions are routinely administered to preterm infants with thrombocytopenia to prevent bleeding. The incidence of thrombocytopenia and administration of platelet transfusion are both inversely related to the gestational age at birth. Currently, there is uncertainty regarding the optimal platelet transfusion threshold, particularly among the most immature infants in the first week of life, which represents the period of highest bleeding risk.

The NeoPlaTT trial was designed to address this pressing uncertainty in the highest risk population (<27 weeks GA). It will test whether a threshold of 20x10^9/L could be safely used after the first week of life, when the risk of serious bleeding is significantly lower, and reduce the need for platelet transfusion altogether. The results of this study have a potential to change clinical practice and improve outcomes in this vulnerable population, while also decreasing costs and resource utilization.

This is a randomized trial with 1:1 allocation to parallel arms. Infants, inborn or outborn, who are admitted to participating NICUs, and who meet the inclusion and exclusion criteria, will be invited to enroll into the trial for platelet count monitoring. Only consented and enrolled infants meeting the additional platelet count trigger of < 50 x 10^9/L (postnatal days 1-7) or <35 x 10^9/L (8 or more postnatal days) will be randomized. Postnatal day 1 starts at birth. Randomization will be allowed to occur up to 36 6/7 weeks' PMA; subjects will be monitored through 40 0/7 weeks PMA. Approximately 30% of consented and enrolled infants are expected to meet the platelet count threshold for randomization.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 23 0/7 to 26 6/7 weeks
* Postnatal age of < 48 hours

Exclusion Criteria:

* Comfort care or withdrawal of care planned
* Neonatal alloimmune thrombocytopenia or suspected/confirmed congenital platelet or bleeding disorder
* Receipt of platelet transfusion
* No receipt of Vitamin K
* Parents/guardian decline consent

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2433 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Survival without major or severe bleeding | Randomization to 40 0/7 weeks postmenstrual age, death, discharge, or transfer outside of the Study Center, whichever occurs first (an average of 98 days postnatal age)
  Bleeding will be assessed using the neonatal Bleeding Assessment Tool (NeoBAT), a validated bleeding assessment tool (Venkatesh V, 2013)

SECONDARY OUTCOMES:
Death | Randomization to 52 0/7 weeks' postmenstrual age, death, discharge, or transfer outside of the Study Center, whichever occurs first, per Neonatal Research Network Generic Research Database Registry protocol.
Major or severe bleeding | Randomization to 40 0/7 weeks postmenstrual age, death, discharge, or transfer outside of the Study Center, whichever occurs first (an average of 98 days postnatal age)
  Bleeding will be assessed using the neonatal Bleeding Assessment Tool (NeoBAT), a validated bleeding assessment tool (Venkatesh V, 2013)
Number of platelet transfusions | Randomization to 40 0/7 weeks postmenstrual age, death, discharge, or transfer outside of the Study Center, whichever occurs first (an average of 98 days postnatal age)
At least one platelet transfusion | Randomization to 40 0/7 weeks postmenstrual age, death, discharge, or transfer outside of the Study Center, whichever occurs first (an average of 98 days postnatal age)
Bronchopulmonary dysplasia among survivors to 36 weeks postmenstrual age | At 36 weeks postmenstrual age
Retinopathy of Prematurity (ROP) | Randomization to 52 0/7 weeks' postmenstrual age, death, discharge, or transfer outside of the Study Center, whichever occurs first, per Neonatal Research Network Generic Research Database Registry protocol.
  Stage 3 ROP, or stage 1 or 2 in Zone 1, or plus disease
Periventricular leukomalacia | Randomization to 52 0/7 weeks' postmenstrual age, death, discharge, or transfer outside of the Study Center, whichever occurs first, per Neonatal Research Network Generic Research Database Registry protocol.

OTHER OUTCOMES:
Late-onset sepsis | Randomization to 40 0/7 weeks postmenstrual age, death, discharge, or transfer outside of the Study Center, whichever occurs first (an average of 98 days postnatal age)
Necrotizing enterocolitis | Randomization to 40 0/7 weeks postmenstrual age, death, discharge, or transfer outside of the Study Center, whichever occurs first (an average of 98 days postnatal age)
  Modified Bells Stage IIA or greater
Thrombosis requiring therapy | Randomization to 40 0/7 weeks postmenstrual age, death, discharge, or transfer outside of the Study Center, whichever occurs first (an average of 98 days postnatal age)
  Thrombosis requiring therapy such as heparin, enoxaparin, or aspirin

CONTACTS AND LOCATIONS:
Overall Officials: Ravi M Patel, MD, Principal Investigator — Emory University
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - University of Colorado, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Northwestern Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Pediatrix Medical Group, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. The NRN plans to share de-identified data after final publication in an NIH supported data repository such as the NICHD Data and Specimen Hub (https://dash.nichd.nih.gov).

REFERENCES:
- [Background] Venkatesh V, Curley A, Khan R, Clarke P, Watts T, Josephson C, Muthukumar P, New H, Seeney F, Morris S, Stanworth S. A novel approach to standardised recording of bleeding in a high risk neonatal population. Arch Dis Child Fetal Neonatal Ed. 2013 May;98(3):F260-3. doi: 10.1136/archdischild-2012-302443. Epub 2012 Nov 9. PMID 23144007